CLINICAL TRIAL: NCT00037037
Title: A Phase I Study of Peptide Based Vaccine Therapy in Patients With High-Risk or Metastatic Melanoma
Brief Title: Vaccine Therapy With or Without Sargramostim in Treating Patients With High-Risk or Metastatic Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069357; CPMC-IRB-13824; LUDWIG-LUD00-025; NCI-G02-2068
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2004-05

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — MART-1 Antigen; sargramostim

INTERVENTIONS:
Biological: MAGE-10.A2
Biological: MART-1 antigen
Biological: NY-ESO-1 peptide vaccine
Biological: sargramostim
Biological: tyrosinase peptide

SUMMARY:
RATIONALE: Vaccines made from peptides may make the body build an immune response to kill tumor cells. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood. Combining vaccine therapy with sargramostim may kill more tumor cells.

PURPOSE: Randomized phase I trial to study the effectiveness of vaccine therapy with or without sargramostim in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the safety of melanoma peptide vaccine with or without sargramostim (GM-CSF) in patients with high-risk or metastatic melanoma.
* Compare changes in peptide-specific cellular and humoral immunologic profiles in patients treated with these regimens.
* Compare tumor response in patients treated with these regimens.

OUTLINE: This is a randomized, open-label study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive melanoma peptide vaccine comprising tyrosinase leader injected at 2 separate sites, Melan-A ELA injected at another site, NY-ESO-1a and NY-ESO-1b combined and injected at one site, and MAGE-10.A2 injected at another site, intradermally once weekly on weeks 1-6.
* Arm II: Patients receive vaccine as in arm I. Patients also receive sargramostim (GM-CSF) subcutaneously daily beginning 2 days before each vaccination and continuing for 5 days.

Treatment in both arms continues through week 6 in the absence of disease progression or unacceptable toxicity.

Patients are followed at 2 weeks.

PROJECTED ACCRUAL: A total of 20 patients (10 per treatment arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed high-risk stage III or IV melanoma

  * Stage III disease less than 6 months after surgical resection

    * Completed prior interferon alfa therapy OR
    * Progressive disease or major adverse events during prior interferon alfa therapy
  * Stage III disease at least 6 months after surgical resection

    * Declined, failed, or completed prior standard therapy
  * Stage IV disease

    * Declined, failed, or completed prior standard therapy
* HLA-A2 positive
* No CNS metastases unless treated and stable

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 80-100%

Life expectancy:

* At least 4 months

Hematopoietic:

* Neutrophil count at least 1,500/mm3
* Lymphocyte count at least 500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 9.0 g/dL (10.0 g/dL if less than 50 kg)
* No bleeding disorder

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* No hepatitis B or C positivity

Renal:

* Creatinine no greater than 1.8 mg/dL

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* HIV negative
* No other serious illness
* No serious infection requiring antibiotics
* No history of immunodeficiency disease or autoimmune disease
* No psychiatric or addictive disorder that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior bone marrow or stem cell transplantation
* At least 4 weeks since prior immunotherapy or biologic therapy
* No other concurrent immunotherapy or biologic therapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No concurrent chemotherapy

Endocrine therapy:

* No concurrent systemic corticosteroids
* No concurrent steroids except topical or inhalational steroids
* Concurrent hormonal therapy allowed

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior surgery

Other:

* At least 4 weeks since prior investigational agents
* Concurrent noncytotoxic anticancer therapy allowed
* No concurrent immunosuppressive therapy
* No concurrent antihistamines
* No concurrent non-steroidal anti-inflammatory drugs except in low doses for prevention of an acute cardiovascular event or pain control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos P. Papadopoulos, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York, United States